CLINICAL TRIAL: NCT01175187
Title: Intrapartum Fever and Histopathological Placental Findings
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: ob&anesth Unit, wolfson medical center
Other Study IDs: 1077
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Histological Placental Inflamation With or Without Fever
Keywords: evron

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: degree and location of inflamation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- EPIDURAL FEVER
- EPIDURAL WITHOUT FEVER
- GROUP 1: EPIDURAL FEVER . GROUP 2 EPIDURAL WITHOUT FEVER

SUMMARY:
Intrapartum fever associated with epidural anesthesia is caused by non infectious causes therefore without histological findings

ELIGIBILITY:
Inclusion Criteria:epidural with and without fever

-

Exclusion Criteria:

* Patients with infectious backgroud or prilinged PROM

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 200 normal deliveries
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: shmuel evron, md, Principal Investigator — Tel Aviv University